CLINICAL TRIAL: NCT05392764
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of Empagliflozin in Patients With Acute Heart Failure
Brief Title: Early Treatment With a Sodium-glucose Co-transporter 2 Inhibitor in High-risk Patients With Acute Heart Failure
Acronym: EMPA-AHF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Juntendo University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Yuya Matsue, Associate Professor, Juntendo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: jRCTs031210682
Record Dates: First submitted 2022-05-14; First posted 2022-05-26 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental): Patients will be randomized 1:1 to either empagliflozin or placebo.
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): Placebo matching empagliflozin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — once-daily oral empagliflozin 10 mg
  Arms: Empagliflozin
Drug: Placebo — Placebo matching empagliflozin 10 mg
  Arms: Placebo

SUMMARY:
The EMPA-AHF trial is a multicentre, randomized, double-blind, placebo-controlled trial designed to evaluate the efficacy and safety of early initiation of once-daily oral empagliflozin 10 mg in patients hospitalized for patients with acute heart failure (AHF) who are at a high risk of adverse events.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the below inclusion criteria will be randomized within 12 h after presentation to the hospital

1. Age of ≥20 and <90 years
2. Hospitalized with a diagnosis of acute heart failure, requiring intravenous loop diuretic therapy, and with all of the following characteristics:

   i. Dyspnoea at rest or induced by slight exertion ii. At least two of the following findings: jugular venous distention, pulmonary rales, lower leg edema, and pulmonary congestion on chest X-ray iii. If the patient has a sinus rhythm at the time of admission, BNP ≥350 pg/mL or NT-proBNP ≥1400 pg/mL; if the patient has atrial fibrillation at the time of admission, BNP ≥500 pg/mL or NT-proBNP ≥2000 pg/mL. For patients taking an angiotensin receptor neprilysin inhibitor, only the reference value for NT-proBNP will be applicable.
3. At least one of the following characteristics:

   i. eGFR <60 mL/min/1.73m2, as calculated using the CKD Epidemiology Collaboration for JapaneseModification of Diet in Renal Disease formula ii. Already taking ≥40 mg of oral furosemide during the period before hospitalization. For patients on loop diuretics other than furosemide, the following conversion should be used: oral furosemide 20 mg = oral azosemide 30 mg = oral torasemide 5 mg.

   iii. Urine output of <300 mL during the 2 h following an appropriate dose of intravenous furosemide administered after hospitalization. An appropriate dose of intravenous furosemide is 20 mg for patients who have not been taking furosemide regularly before hospitalization and is the same as, or greater than, the daily oral dose for patients who have been taking furosemide regularly before hospitalization.
4. Provided written consent to participate in the study

Exclusion Criteria:

1. eGFR <20 mL/min/1.73m2 at the time of admission
2. Already taking an SGLT2i within 3 months prior to hospitalization
3. Type 1 diabetes mellitus
4. Systolic blood pressure <90 mmHg
5. Expected to newly require treatment with thiazide, tolvaptan, or carperitide within 48 hours of study drug administration
6. Main cause of acute heart failure hospitalization is not fluid retention (e.g., persistent ventricular tachycardia, persistent atrial fibrillation/atrial flutter with a ventricular response rate of ≥130 bpm, persistent bradycardia with a ventricular response rate of <45 bpm, an infection, severe anemia, and an acute exacerbation of COPD)
7. Acute coronary syndrome, pulmonary thromboembolism, or a cerebrovascular accident is the main cause of the present hospitalization.
8. At risk of ketoacidosis or hyperosmolar hyperglycaemia
9. On dialysis, including peritoneal dialysis, or the initiation of dialysis during hospitalization is planned
10. Pregnant or lactating women
11. Underwent the following therapeutic interventions within 30 days: cardiovascular surgery (e.g., coronary artery bypass grafting, surgery for valvular heart disease, transcatheter aortic valve implantation, percutaneous coronary intervention, percutaneous edge-to-edge mitral valve repair, and other types of surgery at the investigator's discretion) and implantation of an implantable defibrillator, cardiac resynchronization therapy defibrillator, or implantable ventricular-assist device
12. A diagnosis of acute coronary syndrome, cerebral infarction, or transient ischemic attack made within 90 days
13. Ventricular tachycardia with syncope within 90 days
14. Heart transplant recipient or listed for heart transplantation and expected to undergo transplantation during the present treatment; implanted with an implantable ventricular-assist device or expected to require an implantable ventricular-assist device during the present treatment; or expected to switch to palliative care
15. Intubated at the time of screening or expected to require intubation within within 48 hours of study drug administration
16. Severe valvular heart disease expected to be treated with thoracostomy or catheterization (a reason to exclude secondary mitral or tricuspid regurgitation due to reduced cardiac function does not exist, except for the absence of a plan to perform cardiac surgery or therapeutic catheterization)
17. A diagnosis of secondary cardiomyopathy such as amyloidosis, cardiac sarcoidosis, hemochromatosis, Fabry disease, and muscular dystrophy. Heart failure due to takotsubo cardiomyopathy, obstructive hypertrophic cardiomyopathy, complex congenital heart disease (as determined by the investigator), or pericardial constriction.
18. A diagnosis of peripartum cardiomyopathy made within 6 months
19. Active myocarditis
20. Presence of uncontrolled thyroid disease
21. Acute cardiac structural abnormalities (e.g., acute mitral regurgitation due to ruptured chordae tendineae)
22. Symptomatic bradycardia or complete atrioventricular block, being treated with a temporary pacemaker implantation at the time of admission, or expected to require a temporary pacemaker implantation in the future. Patients who have already been treated with a permanent pacemaker implantation do not meet the exclusion criteria.
23. Serious liver disorder (an increase in AST, ALT, or ALP level ≥3 times the upper limit of normal) or cirrhosis with varices or other findings suggestive of portal hypertension
24. Alcohol use disorder of at least mild severity according to the DSM-V
25. A diagnosis of active malignancy or suspected active malignancy made within 2 years
26. Coexisting diseases other than heart failure with an expected survival prognosis of ≤1 year
27. Participation in a clinical study of another drug 30 days before hospitalization
28. Patients considered to require fasting at screening.
29. Other conditions likely to interfere with the patient's safety or compliance with the protocol
30. Other patients who are considered unsuitable by the principal investigator or other investigators

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
A hierarchical composite endpoint consisting of death within 90 days, heart failure rehospitalization within 90 days, WHF during hospitalization, and urine output up to 48 hours after treatment initiation, assessed by the win ratio | Up to 90 days
  WHF, worsening heart failure

SECONDARY OUTCOMES:
A hierarchical composite endpoint consisting of death within 90 days, heart failure readmission within 90 days, and WHF during hospitalization | Up to 90 days
  WHF, worsening heart failure
A composite endpoint consisting of WHF during hospitalization, death, heart failure rehospitalization, urgent visit for WHF, intensification of diuretic therapy, and worsening NYHA class within 90 days | Up to 90 days
  WHF, worsening heart failure
Change in NT-proBNP from randomization to 48 hours | Evaluated at 48 hours after randomization
Diuretic response, calculated as urine output achieved by loop diuretics (40 mg intravenous furosemide-equivalent dose) at 48 h after treatment initiation | Evaluated at 48 hours after randomization
Improvement in KCCQ-TSS of ≥5 points from randomization to 30 and 90 days after treatment initiation | Up to 90 days
  KCCQ-TSS, Kansas City Cardiomyopathy Questionnaire - Total Symptom Score. The scores range from 0 to 100, with 100 being the best possible score.
Time to hemodynamic stabilization during index hospitalization | During index hospitalization
Re-worsening of heart failure during index hospitalization | During index hospitalization
Heart failure rehospitalization | Up to 90 days
Death | Up to 90 days
Urine output during the 48 h after randomization | Evaluated at 48 hours after randomization
Cardiovascular death | Up to 90 days
Change in the visual analog scale score for dyspnea from after randomization to 24 and 48 h | Evaluated at 24 and 48 hours after randomization
  The scores range from 0 to 100, with 100 being the best possible score.
Change in high sensitivity cardiac troponin T | Evaluated at 48 hours after randomization
Change in the KCCQ-TSS after randomization to 30 and 90 days | Up to 90 days
  KCCQ-TSS, Kansas City Cardiomyopathy Questionnaire - Total Symptom Score. The scores range from 0 to 100, with 100 being the best possible score.
Composite of renal replacement therapy, renal transplantation, eGFR <15 mL/min/1.73m2, ≥50% decrease in eGFR compared to the first sample or a ≥2-fold increase in creatinine level compared to the first sample within 90 days of randomization | Up to 90 days
Trend in eGFR after randomization to 24 h, 48 h, 30 days, and 90 days | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Yuya Matsue, MD, Principal Investigator — Department of Cardiovascular Biology and Medicine, Juntendo University Graduate School of Medicine
Locations (61):
- Japan (61):
  - Anjo Kosei Hospital, Anjo, Aichi-ken
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Hyogo Prefectural Awaji Medical Center, Sumoto, Awaji
  - Funabashi Municipal Medical Center, Funabashi, Chiba
  - Kameda Medical Center, Kamogawa, Chiba
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Fukuokaken Saiseikai Futsukaichi Hospital, Chikushino-shi, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - Kushiro-sanjikai Hospital, Kushiro, Hokkaido
  - Medical Corporation Sapporo Heart Center, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Tsuchiura Kyodo General Hospital, Tsuchiura, Ibaraki
  - Iwate Prefectural Cyuou Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - St.Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Nara Medical University Hospital, Kashihara, Nara
  - Urasoe General Hospital, Urasoe, Okinawa
  - Kindai University Hospital, Sayama, Osaka
  - National Cerebral and Cardiovascular Center Hospital, Suita, Osaka
  - Kasukabe Chuo General Hospital, Kasukabe, Saitama
  - Saitama Medical Center, Kawagoe, Saitama
  - Kawaguchi Cardiovascular and Respiratory Hospital, Kawaguchi, Saitama
  - Soka City Hospital, Sōka, Saitama
  - Seirei Mikatahara General Hospital, Hamamatsu, Shizuoka
  - Juntendo University Shizuoka Hospital, Izunokuni, Shizuoka
  - Saiseikai Utsunomiya Hospital, Utsunomiya, Tochigi
  - Nishiarai Hospital, Adachi City, Tokyo
  - Mitsui Memorial Hospital, Chiyoda City, Tokyo
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - International University of Health and Welfare Mita Hospital, Minato, Tokyo
  - Toranomon Hospital, Minato, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku, Tokyo
  - National Disaster Medical Center, Tachikawa, Tokyo
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Gifu University Graduate school of Medicine, Gifu
  - Hiroshima City Hospital, Hiroshima
  - Kitasato University Hospital, Kanagawa
  - Chikamori Hospital, Kochi
  - Nara Prefecture General Medical Center, Nara
  - Sakakibara Heart Institute of Okayama, Okayama
  - Nakagami Hospital, Okinawa
  - Kitano Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Saitama Citizens Medical Center, Saitama
  - Tokushima University Hospital, Tokushima
  - Juntendo University Hospital, Tokyo
  - Juntendo University Nerima Hospital, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - St. Luke's International Hospital, Tokyo
  - Tokyo General Hospital, Tokyo
  - Tokyo Medical University, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Tokyo
  - Yokohama City University Medical Center, Yokohama

IPD SHARING:
Plan to Share IPD: Undecided